CLINICAL TRIAL: NCT04271189
Title: A Prospective, Randomized, Parallel-group, Adaptive Design Phase IIb/III, Multicenter Study, to Assess the Efficacy of Polychemotherapy for Inducing Remission of Newly Diagnosed Type 2 Diabetes.
Brief Title: Managing DIabetes Remission After Combined Therapy in EarLy Stage of DiabetEs
Acronym: MIRACLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria di Parma (Other)
Responsible Party: Principal Investigator, Riccardo Bonadonna, Director of Endocrinology Unit, Azienda Ospedaliero-Universitaria di Parma
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-833-12
Record Dates: First submitted 2019-10-15; First posted 2020-02-17 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Newly Diagnosed Type 2 Diabetes
Keywords: Type 2 diabetes; Polychemotherapy; Diabetes remission
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Multicenter, open label pragmatic phase IIb/III RCT with a duration of 3 years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- POLYCHEM (Experimental): Metformin (extended release), Pioglitazone, Sitagliptin and Empaglifozin.
  Interventions: Drug: Metformin-Sitagliptin-Empaglifozin-Pioglitazone
- STANDARD CARE (Active Comparator): Standard of care according to the local health service.
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Metformin-Sitagliptin-Empaglifozin-Pioglitazone — 1000 mg metformin (extended release) b.i.d., pioglitazone 15 mg b.i.d., sitagliptin 100 mg q.d., empaglifozin 10 mg q.d..
  Other Names: POLYCHEM
  Arms: POLYCHEM
Drug: Standard of care — Usual medical care to treat diabetes.
  Other Names: SDC
  Arms: STANDARD CARE

SUMMARY:
Epidemiologic, social and economic burdens of type 2 diabetes mellitus (T2DM) keep rising worldwide. Implementation of T2DM preventive trategies is lagging behind. Metabolic surgery, very low calorie diet can induce T2DM remission, but so far for few patients. The investigators will assess the efficacy to cause T2DM remission (primary end point) and direct costs to the National Health System of a 4-month polychemotherapy (metformin+pioglitazone+sitagliptin+empagliflozin) regimen vs standard care in patients with newly diagnosed T2DM by an open label, pragmatic RCT. Mechanisms of action will be investigated in a sub-cohort by a prolonged OGTT plus dual tracer technique and modeling of beta cell function.

If proved efficacious in this proof-of-concept study and inducer of durable remission in the future, T2DM polychemotherapy will turn out to be a convenient, relatively unexpensive strategy to restrain prevalence of T2DM and its complications and to alleviate its personal, social and economic burden.

DETAILED DESCRIPTION:
Hypothesis: at diagnosis of T2DM, a 4 month course of oral polychemotherapy (POLYCHEM), by engaging multiple glucose lowering mechanisms, results into euglycemia and, after suspension, in T2DM remission in a clinically significant higher number of patients when compared to standard diabetes care (SDC).

* Diabetes remission: simultaneous nondiabetic values of fasting glucose, 2-hour glucose (after OGTT) and HbA1c for at least 12 months with no pharmacologic/surgical treatment of diabetes.
* Complete remission: all values of fasting glucose, 2-hour glucose and HbA1c are within the limits of normal glucose regulation; otherwise, remission is partial.
* Hyperglycemia remission as in diabetes remission, but duration<12 months.

Based on the "Consensus Report: Definition and Interpretation of Remission in Type 2 Diabetes" published on Diabetes Care 2021;44(10):2438-2444, remission should be defined as a return of HbA1c to <6.5% (<48 mmol/mol) that occurs spontaneously or following an intervention and that persists for at least 3 months in the absence of usual glucose-lowering pharmacotherapy.

A POLYCHEM (metformin, pioglitazone, sitagliptin and empagliflozin) will be used to improve:

1. Insulin sensitivity of endogenous glucose output (EGO) and peripheral (muscle) glucose uptake (PGU);
2. Beta cell function;
3. GLP-1 and GIP bioavailability. To these effects, the direct glycosuric action of EMPA is added; EMPA effects on alpha cell and liver (increased glucagon secretion and EGO), may be, at least in part, counterbalanced by SITA and MET/PIO, respectively. Increased heart failure events with PIO may be, at least in part, counteracted by EMPA.

In many patients POLYCHEM should result in stable euglycemia, with negligible risk of hypoglycemia, and the number of patients in T2DM remission should be much higher than with MET+SU. The underpinning is that euglycemia reverses the detrimental effects of glucose toxicity and glucose regulation can be maintained in the nondiabetic range.

If the invesigators hypothesis is proved, POLYCHEM would be a convenient, simple and relatively unexpensive strategy to induce remission in a great number of patients with newly diagnosed T2DM. Novel, more efficacious goals of therapy could be introduced. Duration of remission is expected to delay the processes which result into the T2DM related risk of tissue damage. At the patient acceptance level, the trade off between the full T2DM burden (diabetes, its care and the risk of its complications) and the risk of T2DM relapse should favor the latter. At the society level, achieving a durable remission in a substantial number of these patients should attenuate, or even annull, the rises in prevalence, burden and tolls of "active" T2DM.

Patients with newly diagnosed (i.e. less than 6 months) T2DM will be recruited in the Diabetes Outpatient Clinics and will provide informed written consent before participation. After a screening visit (V0), patients will be randomized 1:1, with center stratification through web-based data collection (eCRF), to receive POLYCHEM or SDC with standard lifestyle intervention in both.

In both arms, patients will undergo planned visits at week 0 (V1), week 16 (V2), and week 28 (V3), after at least 3 days of drug washout. Patients will perform weekly a 6-point home blood glucose profile. Between week 17 and week 28, if a patient in hyperglycemia remission relapses, V3 will be anticipated (V3B), after which the patient will be treated as in SDC and will be re-evaluated at week 28 .

Visit procedures:

* V0: assessment of patient eligibility , including medical history, physical examination, and lab exams, if needed.
* V0S: between V0 and V1; signature of informed written consent and randomization.
* V1, V2, V3 and V3B: assessment of anthropometry, ambulatory blood pressure and heart rate, WBC, fasting glucose, HbA1c, lipids, AST, ALT, creatinine, lipase, urine analysis, microalbuminuria, insulin, C-peptide, glucagon, GLP-1, GIP, quality of life (QoL), and, only in V1, blood for DNA collection (the last for post hoc studies).

POLYCHEM-ARM: After V1, patients will start POLYCHEM (MET titrated to 1000 mg b.i.d., PIO 15 mg b.i.d., SITA 100 mg q.d., EMPA 10 mg q.d.) for 16 weeks, at the end of which (V2) patients in hyperglycemia remission stop drug therapy, the others are transferred to SDC. Patients with MET intolerance will be treated with PIO+SITA+EMPA only.

SDC-ARM: After V1, patients will continue their SDC for 16 weeks, at the end of which (V2) patients in hyperglycemia remission stop drug therapy, the others continue SDC.

ELIGIBILITY:
Inclusion criteria:

* Age 35-75 years;
* HbA1c <= 10.0% (86 mmol/mol);
* T2DM diagnosis (< 6 months)
* BMI>=23 and <=40 kg/m2
* Fasting C-peptide > 0.3 nmol/l;
* GAD-antibody negative.

Exclusion criteria:

* Diagnosis of type 1 diabetes;
* History of cancer in the previous 5 years;
* Multiple daily insulin treatment;
* Acute cardiovascular event within the previous 6 months;
* Chronic heart failure;
* eGFR < 45 ml.min-1.1.73 m2 according to the MDRD formula;
* Women of child bearing potential with no use of acceptable contraception;
* Presence of diabetic retinopathy;
* Contraindications to the use of any drug of POLYCHEM.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Assess the T2DM remission rate in patients with newly diagnosed T2DM treated with either POLYCHEM or with SDC for 16 weeks. | 12 weeks after the end of treatment
  Remission was defined as HbA1c <6.5% or 48mmol/mol for at least 12 weeks without pharmacologic or surgical treatment for diabetes.

SECONDARY OUTCOMES:
Assess the proportion of complete T2DM remission rate in the 2 groups | 12 weeks after the end of treatment
  Normal measures of glucose metabolism (fasting glucose and HbA1c in normal range), for at least 12weeks without pharmacologic or surgical treatment for diabetes.
Monitor the quality of life EQ-5D-DL | 0, 16, 28 weeks
  Will be monitored through EQ-5D-DL questionnaires.
Monitor the quality of life ADDQOL | 0, 16, 28 weeks
  QoL will be monitored through ADDQOL questionnaires.
Monitor the costs of National Health System service utilization | 0, 16, 28 weeks
  All accesses to the National Healthcare System resources by each patient (visits, treatments, supplies, hospital admissions, etc.) will be retrieved from the Regional Health Registries and recorded. Costs will be assessed from a public purchaser perspective. For this reason all costs will refer to the reimbursement provided to the health facilities by the national health system.
Quantify the effects of either POLYCHEM or SDC on the main determinants of glucose regulation | 0, 16, 28 weeks
  In all patients C-peptide will be used to compute static surrogate indexes of insulin sensitivity and beta cell function.
Quantify the effects of either POLYCHEM or SDC on the main determinants of glucose regulation | 0, 16, 28 weeks
  In all patients insulin values will be used to compute static surrogate indexes of insulin sensitivity and beta cell function.
Quantify the effects of either POLYCHEM or SDC on the main determinants of glucose regulation | 0, 16, 28 weeks
  Glucagon values will provide indexes of alpha cell function and of gut K- and L-cell function. Their role in predicting and/or explaining T2DM remission and/or relapse will be assessed.
Quantify the effects of either POLYCHEM or SDC on the main determinants of glucose regulation | 0, 16, 28 weeks
  GLP-1 values will provide indexes of alpha cell function and of gut K- and L-cell function. Their role in predicting and/or explaining T2DM remission and/or relapse will be assessed.
Quantify the effects of either POLYCHEM or SDC on the main determinants of glucose regulation | 0, 16, 28 weeks
  GIP values will provide indexes of alpha cell function and of gut K- and L-cell function. Their role in predicting and/or explaining T2DM remission and/or relapse will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Bonadonna, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma
Locations (1):
- Azienda Ospedaliero Universitaria di Parma, Parma, Parma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gregg EW, Li Y, Wang J, Burrows NR, Ali MK, Rolka D, Williams DE, Geiss L. Changes in diabetes-related complications in the United States, 1990-2010. N Engl J Med. 2014 Apr 17;370(16):1514-23. doi: 10.1056/NEJMoa1310799. PMID 24738668
- [Background] American Diabetes Association. 4. Prevention or Delay of Type 2 Diabetes. Diabetes Care. 2016 Jan;39 Suppl 1:S36-8. doi: 10.2337/dc16-S007. No abstract available. PMID 26696678
- [Background] Alouki K, Delisle H, Bermudez-Tamayo C, Johri M. Lifestyle Interventions to Prevent Type 2 Diabetes: A Systematic Review of Economic Evaluation Studies. J Diabetes Res. 2016;2016:2159890. doi: 10.1155/2016/2159890. Epub 2016 Jan 13. PMID 26885527
- [Background] Aziz Z, Absetz P, Oldroyd J, Pronk NP, Oldenburg B. A systematic review of real-world diabetes prevention programs: learnings from the last 15 years. Implement Sci. 2015 Dec 15;10:172. doi: 10.1186/s13012-015-0354-6. PMID 26670418
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Li G, Zhang P, Wang J, Gregg EW, Yang W, Gong Q, Li H, Li H, Jiang Y, An Y, Shuai Y, Zhang B, Zhang J, Thompson TJ, Gerzoff RB, Roglic G, Hu Y, Bennett PH. The long-term effect of lifestyle interventions to prevent diabetes in the China Da Qing Diabetes Prevention Study: a 20-year follow-up study. Lancet. 2008 May 24;371(9626):1783-9. doi: 10.1016/S0140-6736(08)60766-7. PMID 18502303
- [Background] DeFronzo RA, Tripathy D, Schwenke DC, Banerji M, Bray GA, Buchanan TA, Clement SC, Henry RR, Hodis HN, Kitabchi AE, Mack WJ, Mudaliar S, Ratner RE, Williams K, Stentz FB, Musi N, Reaven PD; ACT NOW Study. Pioglitazone for diabetes prevention in impaired glucose tolerance. N Engl J Med. 2011 Mar 24;364(12):1104-15. doi: 10.1056/NEJMoa1010949. PMID 21428766
- [Background] Carlsson LM, Peltonen M, Ahlin S, Anveden A, Bouchard C, Carlsson B, Jacobson P, Lonroth H, Maglio C, Naslund I, Pirazzi C, Romeo S, Sjoholm K, Sjostrom E, Wedel H, Svensson PA, Sjostrom L. Bariatric surgery and prevention of type 2 diabetes in Swedish obese subjects. N Engl J Med. 2012 Aug 23;367(8):695-704. doi: 10.1056/NEJMoa1112082. PMID 22913680
- [Background] Schauer PR, Mingrone G, Ikramuddin S, Wolfe B. Clinical Outcomes of Metabolic Surgery: Efficacy of Glycemic Control, Weight Loss, and Remission of Diabetes. Diabetes Care. 2016 Jun;39(6):902-11. doi: 10.2337/dc16-0382. PMID 27222548
- [Background] Lim EL, Hollingsworth KG, Aribisala BS, Chen MJ, Mathers JC, Taylor R. Reversal of type 2 diabetes: normalisation of beta cell function in association with decreased pancreas and liver triacylglycerol. Diabetologia. 2011 Oct;54(10):2506-14. doi: 10.1007/s00125-011-2204-7. Epub 2011 Jun 9. PMID 21656330
- [Background] Sattar N. Revisiting the links between glycaemia, diabetes and cardiovascular disease. Diabetologia. 2013 Apr;56(4):686-95. doi: 10.1007/s00125-012-2817-5. Epub 2013 Jan 27. PMID 23354123
- [Background] Buse JB, Caprio S, Cefalu WT, Ceriello A, Del Prato S, Inzucchi SE, McLaughlin S, Phillips GL 2nd, Robertson RP, Rubino F, Kahn R, Kirkman MS. How do we define cure of diabetes? Diabetes Care. 2009 Nov;32(11):2133-5. doi: 10.2337/dc09-9036. No abstract available. PMID 19875608
- [Background] Weng J, Li Y, Xu W, Shi L, Zhang Q, Zhu D, Hu Y, Zhou Z, Yan X, Tian H, Ran X, Luo Z, Xian J, Yan L, Li F, Zeng L, Chen Y, Yang L, Yan S, Liu J, Li M, Fu Z, Cheng H. Effect of intensive insulin therapy on beta-cell function and glycaemic control in patients with newly diagnosed type 2 diabetes: a multicentre randomised parallel-group trial. Lancet. 2008 May 24;371(9626):1753-60. doi: 10.1016/S0140-6736(08)60762-X. PMID 18502299
- [Background] Sosnowski C, Janeczko-Sosnowska E. [Commentary to the article: Kahn SE, Haffner SM, Heise MA, et al. ADOPT Study Group. Glycemic durability of rosiglitazone, metformin, or glyburide monotherapy. N Engl J Med 2006; 355: 2427-43]. Kardiol Pol. 2007 Feb;65(2):214-6; discussion 216-7. No abstract available. Polish. PMID 17366371
- [Background] Kahn SE, Cooper ME, Del Prato S. Pathophysiology and treatment of type 2 diabetes: perspectives on the past, present, and future. Lancet. 2014 Mar 22;383(9922):1068-83. doi: 10.1016/S0140-6736(13)62154-6. Epub 2013 Dec 3. PMID 24315620
- [Background] Ferrannini E, Muscelli E, Frascerra S, Baldi S, Mari A, Heise T, Broedl UC, Woerle HJ. Metabolic response to sodium-glucose cotransporter 2 inhibition in type 2 diabetic patients. J Clin Invest. 2014 Feb;124(2):499-508. doi: 10.1172/JCI72227. Epub 2014 Jan 27. PMID 24463454
- [Background] Muscelli E, Casolaro A, Gastaldelli A, Mari A, Seghieri G, Astiarraga B, Chen Y, Alba M, Holst J, Ferrannini E. Mechanisms for the antihyperglycemic effect of sitagliptin in patients with type 2 diabetes. J Clin Endocrinol Metab. 2012 Aug;97(8):2818-26. doi: 10.1210/jc.2012-1205. Epub 2012 Jun 8. PMID 22685234
- [Background] Basu R, Shah P, Basu A, Norby B, Dicke B, Chandramouli V, Cohen O, Landau BR, Rizza RA. Comparison of the effects of pioglitazone and metformin on hepatic and extra-hepatic insulin action in people with type 2 diabetes. Diabetes. 2008 Jan;57(1):24-31. doi: 10.2337/db07-0827. Epub 2007 Oct 3. PMID 17914032
- [Background] Dormandy JA, Charbonnel B, Eckland DJ, Erdmann E, Massi-Benedetti M, Moules IK, Skene AM, Tan MH, Lefebvre PJ, Murray GD, Standl E, Wilcox RG, Wilhelmsen L, Betteridge J, Birkeland K, Golay A, Heine RJ, Koranyi L, Laakso M, Mokan M, Norkus A, Pirags V, Podar T, Scheen A, Scherbaum W, Schernthaner G, Schmitz O, Skrha J, Smith U, Taton J; PROactive Investigators. Secondary prevention of macrovascular events in patients with type 2 diabetes in the PROactive Study (PROspective pioglitAzone Clinical Trial In macroVascular Events): a randomised controlled trial. Lancet. 2005 Oct 8;366(9493):1279-89. doi: 10.1016/S0140-6736(05)67528-9. PMID 16214598
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Fonseca V, Staels B, Morgan JD 2nd, Shentu Y, Golm GT, Johnson-Levonas AO, Kaufman KD, Goldstein BJ, Steinberg H. Efficacy and safety of sitagliptin added to ongoing metformin and pioglitazone combination therapy in a randomized, placebo-controlled, 26-week trial in patients with type 2 diabetes. J Diabetes Complications. 2013 Mar-Apr;27(2):177-83. doi: 10.1016/j.jdiacomp.2012.09.007. Epub 2012 Oct 30. PMID 23116881
- [Background] Kovacs CS, Seshiah V, Merker L, Christiansen AV, Roux F, Salsali A, Kim G, Stella P, Woerle HJ, Broedl UC; EMPA-REG EXTEND PIO investigators. Empagliflozin as Add-on Therapy to Pioglitazone With or Without Metformin in Patients With Type 2 Diabetes Mellitus. Clin Ther. 2015 Aug;37(8):1773-88.e1. doi: 10.1016/j.clinthera.2015.05.511. Epub 2015 Jun 29. PMID 26138864
- [Background] Trombetta M, Dauriz M, Bonetti S, Travia D, Boselli L, Santi L, Bonora E, Bonadonna RC. Is common genetic variation at IRS1, ENPP1 and TRIB3 loci associated with cardiometabolic phenotypes in type 2 diabetes? An exploratory analysis of the Verona Newly Diagnosed Type 2 Diabetes Study (VNDS) 5. Nutr Metab Cardiovasc Dis. 2016 Mar;26(3):232-8. doi: 10.1016/j.numecd.2016.01.002. Epub 2016 Jan 14. PMID 26868433
- [Background] Zwarenstein M, Treweek S, Gagnier JJ, Altman DG, Tunis S, Haynes B, Oxman AD, Moher D; CONSORT group; Pragmatic Trials in Healthcare (Practihc) group. Improving the reporting of pragmatic trials: an extension of the CONSORT statement. BMJ. 2008 Nov 11;337:a2390. doi: 10.1136/bmj.a2390. PMID 19001484
- [Background] Apolone G, Mosconi P. The Italian SF-36 Health Survey: translation, validation and norming. J Clin Epidemiol. 1998 Nov;51(11):1025-36. doi: 10.1016/s0895-4356(98)00094-8. PMID 9817120
- [Background] Trento M, Passera P, Borgo E, Tomalino M, Bajardi M, Cavallo F, Porta M. A 5-year randomized controlled study of learning, problem solving ability, and quality of life modifications in people with type 2 diabetes managed by group care. Diabetes Care. 2004 Mar;27(3):670-5. doi: 10.2337/diacare.27.3.670. PMID 14988283
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Bonadonna RC, Heise T, Arbet-Engels C, Kapitza C, Avogaro A, Grimsby J, Zhi J, Grippo JF, Balena R. Piragliatin (RO4389620), a novel glucokinase activator, lowers plasma glucose both in the postabsorptive state and after a glucose challenge in patients with type 2 diabetes mellitus: a mechanistic study. J Clin Endocrinol Metab. 2010 Nov;95(11):5028-36. doi: 10.1210/jc.2010-1041. Epub 2010 Aug 25. PMID 20739378
- [Background] Daniele G, Gaggini M, Comassi M, Bianchi C, Basta G, Dardano A, Miccoli R, Mari A, Gastaldelli A, Del Prato S. Glucose Metabolism in High-Risk Subjects for Type 2 Diabetes Carrying the rs7903146 TCF7L2 Gene Variant. J Clin Endocrinol Metab. 2015 Aug;100(8):E1160-7. doi: 10.1210/jc.2015-1172. Epub 2015 Jun 5. PMID 26046964
- [Background] Nadalini L, Zenti MG, Masotto L, Indelicato L, Fainelli G, Bonora F, Battistoni M, Romani B, Genna M, Zoppini G, Bonora E. Improved quality of life after bariatric surgery in morbidly obese patients. Interdisciplinary group of bariatric surgery of Verona (G.I.C.O.V.). G Chir. 2014 Jul-Aug;35(7-8):161-4. PMID 25174289
- [Background] Riddle MC, Cefalu WT, Evans PH, Gerstein HC, Nauck MA, Oh WK, Rothberg AE, le Roux CW, Rubino F, Schauer P, Taylor R, Twenefour D. Consensus Report: Definition and Interpretation of Remission in Type 2 Diabetes. Diabetes Care. 2021 Aug 30;44(10):2438-44. doi: 10.2337/dci21-0034. Online ahead of print. PMID 34462270